CLINICAL TRIAL: NCT07001293
Title: Supporting Expectant Mothers With ADHD Through the Transition to Parenthood: A Pilot RCT
Brief Title: Expectant Moms Managing Attention-Deficit/ Hyperactivity Disorder
Acronym: MomMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Heather Joseph, Assistant Professor of Psychiatry and Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY25030051
Record Dates: First submitted 2025-04-07; First posted 2025-06-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: ADHD; Perinatal; Behavioral Intervention
Keywords: ADHD; Pregnancy; Perinatal Mental Health; Behavioral Intervention; Parenting; Emotion Regulation; Executive Functioning
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Emotional Regulation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MomMA Intervention (Experimental)
  Interventions: Behavioral: MomMA Intervention
- Treatment As Usual (TAU) (Other): Treatment will be determined by participant and their medical and behavioral health providers.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: MomMA Intervention — The MomMA program is a CBT-based behavioral intervention with components targeted specifically towards expectant parents with ADHD. Treatment will be delivered by therapists embedded in OB care settings.
  Arms: MomMA Intervention
Other: Treatment as Usual (TAU) — Participants will receive treatment as usual, including but not limited to medication and behavioral therapy. No participation in treatment is required.
  Arms: Treatment As Usual (TAU)

SUMMARY:
The goal of this study is to test a behavioral program for pregnant individuals with ADHD. This behavioral program focuses on skills for managing ADHD and related symptoms in pregnancy and postpartum.

This pilot effectiveness-implementation trial aims to (1) preliminarily evaluate the MomMA behavioral intervention compared to treatment as usual (TAU) on clinical outcomes and (2) evaluate implementation outcomes, including feasibility and acceptability of clinic screening within existing OB workflows; assessment and intervention protocols; provider training/fidelity to manual; and all other study protocols from the perspective of real-world providers and participants.

DETAILED DESCRIPTION:
Treating pregnant individuals with ADHD may improve parent and child wellbeing, parent-child interactions, and psychosocial familial factors to enhance family resilience and reduce prevalence/severity of child mental health disorders. The current study will test the MomMA (Moms Managing ADHD) intervention and implement it via a randomized controlled trial (N= 40 pregnant women with ADHD; 20 receiving the behavioral intervention and 20 receiving TAU), delivered by women's health behavioral therapists. Investigators will examine treatment acceptability, feasibility, and appropriateness, as well as implementation factors (fidelity, adherence, facilitators/barriers). In addition, quantitative data will be used to assess parent and child clinical outcomes, including maternal ADHD symptom severity and impairment (primary), parent-child attachment, and infant temperament/behavior. Finally, changes in target mechanisms (executive function and emotion regulation) and whether changes in the target are associated with change in clinical outcomes will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. meets full DSM-5 criteria for ADHD
2. is between 14- and 22-weeks of gestation
3. 18 years of age or older
4. English speaking
5. Lives in Pennsylvania

Exclusion Criteria:

1. substance use disorders requiring dual diagnosis treatment
2. intellectual disability
3. bipolar disorder, psychosis, and major depressive disorder with suicidal ideation
4. the following high complexity medical conditions during pregnancy: maternal cancer, multiples, placenta accreta, and/or fetus known to have a severe congenital condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability | Post Intervention (36 weeks gestational age)
  Therapist and participant report of intervention acceptability will be assessed using the 4-item Acceptability of Intervention Measure (AIM), rated from rated from 1 (completely disagree) to 5 (completely agree).
Intervention Feasibility | Post Intervention (36 weeks gestational age)
  Therapist and participant report of intervention feasibility will be assessed using the 4-item Feasibility of Intervention Measure (FIM), rated from 1 (completely disagree) to 5 (completely agree).
Intervention Appropriateness | Post Intervention (36 weeks gestational age)
  Therapist and participant report of intervention appropriateness will be assessed using the 4-item Intervention Appropriateness Measure (IAM), rated from 1 (completely disagree) to 5 (completely agree).
ADHD Symptom Severity | Post Intervention (36 weeks gestational age) and Postpartum follow-up (4-5 months postpartum)
  Number and severity of ADHD symptoms will be self-reported using the Barkley Adult ADHD Rating Scale-IV (BAARS-IV). Number and severity of ADHD symptoms will be self-reported using the Barkley Adult ADHD Rating Scale-IV (BARRS-IV). Total score (range 18-72) and number of symptoms (0-18) will be determined by summing the Inattention (total score: range 9-36; number of symptoms: range 0-9), Hyperactivity (total score: range 5-20; number of symptoms: range 0-5), and Impulsivity (total score: range 4-16; number of symptoms: range 0-4) subscales. On all scales, higher scores indicate greater ADHD symptoms.
ADHD Functional Impairment | Post Intervention (36 weeks gestational age) and Postpartum follow-up (4-5 months postpartum)
  Impairment in family functioning and self-concept will be assessed on two subscales of the Weiss Functional Impairment Rating Scale (WFIRS-S). Impairment in family functioning and self-concept will be assessed on two subscales of the Weiss Functional Impairment Rating Scale (WFIRS-S). For each scale, mean impairment (range 0-3) and a total impairment score (Family subscale: range 0-24; Self-Concept subscale: range 0-15) will be calculated. Any subscale with at least 2 items scored a 2 or 3, one item scored 3, or a mean score of >1.5 is considered impaired.
Perinatal Mood/Distress | Post Intervention (36 weeks gestational age) and Postpartum follow-up (4-5 months postpartum)
  Symptoms of depression, anxiety, and distress will be assessed using self-report on the Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder scale (GAD-7), and Perceived Stress Scale (PSS). Symptoms of depression, anxiety, and distress will be assessed using self-report on the Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder scale (GAD-7), and Perceived Stress Scale (PSS). The PHQ-9 (total score range 0-27) measures depression, with higher scores indicating greater depressive symptoms. The GAD-7 (total score range 0-21) measures anxiety, with higher scores indicating greater anxiety symptoms. The PSS (total score range 0-40) measures perceived stress, with higher scores indicating greater perceived stress.

SECONDARY OUTCOMES:
Attachment | Postpartum follow-up (4-5 months postpartum)
  Maternal Postnatal Attachment Scale (MPAS) is a 19-item self-report questionnaire, and measures Mother to Baby Attachment during pregnancy. Questions explore maternal interest in and preoccupation with pregnancy, as well as the respondent's emotions towards the growing infant. Similar to the MPAS, each item is equally weighted and has five answer choices, with total scores ranging from 19-95.
Home Environment | Postpartum follow-up (4-5 months postpartum)
  Using the Confusion, Hubbub, and Order Scale, a 15-item self-report scale rated from 1 (Very much like your own home) to 4 (Not at all like your own home). Total scores range from 15-60, with higher scores indicating more chaotic homes.
Infant Behavior | Postpartum follow-up (4-5 months postpartum)
  Infant behavior (temperament and sleep) will be reported by mothers on the Infant Behavior Questionnaire-Short Form (IBQ-R-SF) and the Brief Infant Sleep Questionnaire (BISQ).
Parent-Child Interaction | Postpartum follow-up (4-5 months postpartum)
  Parent affect, warmth, responsiveness, engagement, sensitivity, indifference, intrusiveness, and infant affect, engagement, attentiveness will be rated using the Global Ratings of Mother-Infant Interaction.

OTHER OUTCOMES:
Parent Executive Function | Change from baseline to Post Intervention (36 weeks gestational age)
  Participant will self-report on executive function using the Barkley Deficits in Executive Function Scale (BDEFS). Items are rated from 1 (Never or rarely) to 4 (Very often). Executive Functioning will be assessed as a Target Mechanism. These data will be used in exploratory analyses to determine change from baseline to post-intervention, and whether this change is related to change in clinical outcome measures.
Parent Emotion Regulation | Change from Baseline to Post Intervention (36 weeks gestational age)
  Participant will self-report on executive function using the Difficulties in Emotion Regulation Scale - Short Form (DERS-SF). Items are rated from 1 (Almost never, 0-10%) to 5 (Almost always, 91-100%). Emotion Regulation will be assessed as a Target Mechanism. These data will be used in exploratory analyses to determine change from baseline to post-intervention, and whether this change is related to change in clinical outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Joseph, DO Assistant Professor of Psychiatry and Pediatrics, Principal Investigator — University of Pittsburgh; Andrea Chronis-Tuscano, PhD Joel & Kim Feller Endowed Professor, Principal Investigator — University of Maryland
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial will be shared, after deidentification, via the NIMH National Data Archive.
Time Frame: Data will be shared upon publication or 1 year after the grant end date. Data will be available indefinitely.
URL: https://nda.nih.gov

REFERENCES:
- [Background] Chronis-Tuscano A, Clarke TL, O'Brien KA, Raggi VL, Diaz Y, Mintz AD, Rooney ME, Knight LA, Seymour KE, Thomas SR, Seeley J, Kosty D, Lewinsohn P. Development and preliminary evaluation of an integrated treatment targeting parenting and depressive symptoms in mothers of children with attention-deficit/hyperactivity disorder. J Consult Clin Psychol. 2013 Oct;81(5):918-25. doi: 10.1037/a0032112. Epub 2013 Mar 11. PMID 23477479
- [Background] Joseph HM, Khetarpal SK, Wilson MA, Molina BSG. Parent ADHD Is Associated With Greater Parenting Distress in the First Year Postpartum. J Atten Disord. 2022 Jul;26(9):1257-1268. doi: 10.1177/10870547211066488. Epub 2021 Dec 23. PMID 34937412